CLINICAL TRIAL: NCT01318733
Title: A Multicenter, Open-Label Study to Evaluate the Long-Term Safety and Efficacy of CD07805/47 Gel 0.5% Applied Topically Once Daily for up to 52 Weeks in Subjects With Moderate to Severe Facial Erythema Associated With Rosacea
Brief Title: Study of CD07805/47 Topical Gel in Subjects With Facial Erythema Associated With Rosacea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD.06.SPR.18142
Record Dates: First submitted 2011-03-09; First posted 2011-03-18 (Estimated); Results first posted 2014-01-08 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2014-03

CONDITIONS: Rosacea
Keywords: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CD07805/47 Gel 0.5% (Experimental)
  Interventions: Drug: CD07805/47 gel 0.5%

INTERVENTIONS:
Drug: CD07805/47 gel 0.5% — In this open-label study, all subjects will receive treatment with CD07805/47 gel 0.5% applied once daily, for up to 12 months.

SUMMARY:
A long-term, open-label, non-comparative safety and efficacy study of CD07805/47 gel 0.5% once daily in subjects with moderate to severe facial erythema associated with rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Male or female who is at least 18 years of age or older.
* A clinical diagnosis of facial rosacea.
* A Clinician Erythema Assessment (CEA) score of ≥3 at Screening and at Baseline (prior to study drug application).
* A Patient Self Assessment (PSA) score of ≥3 at Screening and at Baseline (prior to study drug application).

Exclusion Criteria:

* Particular forms of rosacea (rosacea conglobata, rosacea fulminans, isolated rhinophyma, isolated pustulosis of the chin) or other concomitant facial dermatoses that are similar to rosacea such as peri-oral dermatitis, demodicidosis, facial keratosis pilaris, seborrheic dermatitis, acute lupus erythematosus, or actinic telangiectasia.
* Current diagnosis of Raynaud's syndrome, thromboangiitis obliterans, orthostatic hypotension, severe cardiovascular disease, cerebral or coronary insufficiency, renal or hepatic impairment, scleroderma, Sjögren's syndrome, or depression.
* Previous refractive eye surgery such as photorefractive keratectomy (PRK), laser-assisted sub-epithelial keratectomy (LASEK), or laser-assisted in situ keratomileusis (LASIK).
* Current treatment with monoamine oxidase (MAO) inhibitors.
* Current treatment with barbiturates, opiates, sedatives, systemic anesthetics, or alpha-agonists.
* Less than 3 months stable dose treatment with tricyclic anti-depressants, cardiac glycosides, beta blockers or other antihypertensive agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Clark, MD, Principal Investigator — Longmont Clinical PC; Lesly Davidson, MD, Principal Investigator — Palmetto Medical Research; Steven Davis, MD, Principal Investigator — Dermatology Clinical Research Center of San Antonio; Michael Donahue, MD, Principal Investigator — Wilmington Medical Research; Timothy Gardner, MD, Principal Investigator — East Tennessee Medical Research; Michael Gold, MD, Principal Investigator — Tennessee Clinical Research Center; Fasahat Hamzavi, MD, Principal Investigator — Hamzavi Dermatology; Mark Lee, MD, Principal Investigator — Progressive Clinicial Research, PA; Debra Liu, MD, Principal Investigator — Piedmont Medical Research; Keith Loven, MD, Principal Investigator — Rivergate Dermatology Clinical Research Center, PLLC; Michael Maloney, MD, Principal Investigator — Cherry Creek Research, Inc.; Angela Moore, MD, Principal Investigator — Arlington Center for Dermatology; George Murakawa, MD, Principal Investigator — Dermcenter PC - Somerset Skin Centre; Catherine Pointon, MD, Principal Investigator — Metrolina Medical Research; Elyse Rafal, MD, Principal Investigator — DermResearch Center of NewYork, Inc.; Stephen Schleicher, MD, Principal Investigator — DermDox; Joel Schlessinger, MD, Principal Investigator — Skin Specialists, PC; Leonard Swinyer, MD, Principal Investigator — Dermatology Research Center; Amanda Tauscher, MD, Principal Investigator — Compliant Clinical Research; Gary Waterman, MD, Principal Investigator — Deaconess Clinic; Jonathan Weiss, MD, Principal Investigator — Gwinnett Clinical Research Center, Inc.; Morrissa Baskin, MD, Principal Investigator — Wenatchee Valley Medical Center, Clinical Research Department; Steven Kempers, MD, Principal Investigator — Minnesota Clinical Study Center; Ava Shamban, MD, Principal Investigator — The Laser Institute for Dermatology; Harry Sharata, MD, Principal Investigator — Madison Skin & Research, Inc.; Russell Mader, MD, Principal Investigator — TriCities Medical Research; Girish Munavalli, MD, Principal Investigator — Dermatology, Laser & Vein Specialists of the Carolinas
Locations (27):
- United States (27):
  - The Laser Institute for Dermatology, Santa Monica, California
  - Cherry Creek Research, Inc, Denver, Colorado
  - Longmont Clinical PC, Longmont, Colorado
  - Gwinnett Clinical Research Center, Inc, Snellville, Georgia
  - Deaconess Clinic, Evansville, Indiana
  - Compliant Clinical Research, Olathe, Kansas
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Dermcenter PC- Somerset Skin Centre, Troy, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Skin Specialists, PC, Omaha, Nebraska
  - DermResearch Center of New York, Inc, Stony Brook, New York
  - Metrolina Medical Research, Charlotte, North Carolina
  - Dermatology, Laser & Vein Specialists of the Carolinas, Charlotte, North Carolina
  - Wilmington Medical Research, Wilmington, North Carolina
  - Piedmont Medical Research, Winston-Salem, North Carolina
  - DermDox, Hazleton, Pennsylvania
  - Palmetto Medical Research, Mt. Pleasant, South Carolina
  - Rivergate Dermatology Clinical Research Center, PLLC, Goodlettsville, Tennessee
  - East Tennessee Medical Research, Johnson City, Tennessee
  - TriCities Medical Research, Kingsport, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Arlington Center for Dermatology, Arlington, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Progressive Clinical Research, PA, San Antonio, Texas
  - Dermatology Research Center, Salt Lake City, Utah
  - Wenatchee Valley Medical Center - Clinical Research Department, Wenatchee, Washington
  - Madison Skin & Research, Inc., Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- CD07805/47 Gel 0.5%: CD07805/47 Gel 0.5% once daily
Period: Overall Study
Arm/Group | CD07805/47 Gel 0.5%
Started | 449
Completed | 279
Not Completed | 170

BASELINE CHARACTERISTICS:
Arm/Group | CD07805/47 Gel 0.5%
Number analyzed (Participants) | 449
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 395
  >=65 years | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (12.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 336
  Male | 113
Region of Enrollment [Number; unit: participants]
  United States | 449

OUTCOME MEASURES:

1. Primary Outcome: Long Term Safety & Efficacy of CD07805/47 Gel 0.5% in Subjects With Moderate to Severe Facial Erythema Associated With Rosacea.
Description: Static evaluation of erythema severity using the Clinician Erythema Assessment (CEA) - Grade/Description 0 / Clear Skin with no signs of erythema
  1. / Almost clear; slight redness
  2. / Mild erythema; definite redness
  3. / Moderate erythema; marked redness
  4. / Severe erythema; fiery redness
  Change in CEA from Baseline CEA (T0 at Baseline visit Day 1) at T3 of each post-baseline visit, including Day 1.
Time Frame: Over 1 year
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | CD07805/47 Gel 0.5% QD
Number analyzed (Participants) | 449
scores on a scale
  Day 1 / Hour 3 | -1.5 (.88)
  Week 1/ Hour 3 | -1.4 (.85)
  Month 1/ Hour 3 | -1.5 (.83)
  Month 3 / Hour 3 | -1.7 (.84)
  Month 6 / Hour 3 | -1.8 (.88)
  Month 9 / Hour 3 | -1.7 (.9)
  Month 12 / Hour 3 | -1.8 (.83)

ADVERSE EVENTS:
Arm/Group | CD07805/47 Gel 0.5%
Serious Adverse Events (participants affected / at risk) | 12/449
Other Adverse Events (participants affected / at risk) | 101/449
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CD07805/47 Gel 0.5% (N=449)
Abscess tooth w/ secondary submandibular infection (Infections and infestations) | 1 (1)
Osteoarthritis of left hip (Musculoskeletal and connective tissue disorders) | 1 (1)
Advanced squamous cell carcinoma of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Invasive ductal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Distal Esophageal Schatzki's Ring (Gastrointestinal disorders) | 1 (1)
Unstable Angina (Cardiac disorders) | 1 (1)
Right Ovarian Cyst (Reproductive system and breast disorders) | 1 (1)
Sustained Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Atypical Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Synovitis Right Ankle (Musculoskeletal and connective tissue disorders) | 1 (1)
Persistent Abnormal Uterine Bleeding (Reproductive system and breast disorders) | 1 (1)
Bilateral Achilles Tendon ruptures (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CD07805/47 Gel 0.5% (N=449)
Erythema (Skin and subcutaneous tissue disorders) | 35
Rosacea (Skin and subcutaneous tissue disorders) | 24
Flushing (Vascular disorders) | 46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days